CLINICAL TRIAL: NCT03231436
Title: Fixed Dose Versus Height - Adjusted Dose of Intrathecal Hyperbaric Bupivacaine With Opioid for Cesarean Delivery: a Prospective Double-blinded Randomized Trial
Brief Title: Fixed Dose Spinal Bupivacaine for Cesarean Delivery
Acronym: SpinFix-Bupi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartosz Horosz, MD (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor-Investigator, Bartosz Horosz, MD, Principal Investigator, Centre of Postgraduate Medical Education
Organization: Centre of Postgraduate Medical Education (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 65/PB/BHorosz/2017
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Spinal Anesthesia; Cesarean Section
Keywords: intrathecal bupivacaine; hyperbaric bupivacaine; failed spinal
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed dose of 12.5mg bupivacaine (Experimental): Participants that receive the same dose of intrathecal bupivacaine and 25mcg of fentanyl, regardless of their height.
  Interventions: Drug: Fixed dose of 12.5mg bupivacaine
- Height-adjusted dose of bupivacaine (Active Comparator): Participants that receive the dose of intrathecal bupivacaine adjusted to their height and 25mcg of fentanyl
  Interventions: Drug: Height-adjusted dose of bupivacaine

INTERVENTIONS:
Drug: Fixed dose of 12.5mg bupivacaine — Spinal anesthesia performed with 12,5mg of bupivacaine with 25mcg fentanyl for cesarean section
  Arms: Fixed dose of 12.5mg bupivacaine
Drug: Height-adjusted dose of bupivacaine — Spinal anesthesia performed with height-adjusted dose of bupivacaine with 25mcg fentanyl for cesarean section
  Arms: Height-adjusted dose of bupivacaine

SUMMARY:
The study is designed to compare the effectiveness of spinal anesthesia performed with fixed dose of hyperbaric bupivacaine regardless of patient's height and weight and anesthesia with the dose of bupivacaine that is adjusted to their height. Our clinical experience shows that spinal anesthesia using specific, relatively high dose of hyperbaric bupivacaine combined with opioid is very effective, regardless of parturient's weight and height, provides very good surgical conditions and assures patient's comfort while the rate of anesthesia - related complications is similar or less. Therefore, using height-adjusted protocols, although preferred in some centres, might not be necessary in order to provide good anaesthesia for cesarean delivery. Fixed dose regimen may have some additional advantages in obstetric anesthesia settings, as many of cesareans are performed out of hours, giving less room for mistakes in less experienced hands.

Two groups of parturients undergoing cesarean section are to be compared: anesthetized with fixed-dose regimen (intervention group) and anesthetized with height-adjusted dose regimen (control group). Patients are going to be randomized to one of the above groups, two anesthetists will be involved in anesthetic procedure: anesthetist that looks after the patient throughout the procedure will be blinded to the dose of anesthetic given intrathecally. Therefore his judgment of anesthetic effectiveness is not going to be biased and all patients will receive the same perioperative care in terms of fluid therapy, management of possible anesthesia - related complications and postoperative pain control.

Rate of effective spinal anesthetics, defined as adequate block level and no need for additional intraoperative analgesia has been established as primary outcome measure. Secondary outcome measures are rate of complications and amount of opioids used postoperatively. These are going to be statistically compared.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy above 37Hbd scheduled for elective cesarean section
* ASA 1 or 2

Exclusion Criteria:

* absolute contraindications to spinal anesthesia
* delivery in progress
* non-singleton pregnancy
* BMI>35
* ultrasound - based estimation of fetal weight below 10 percentile
* pregnancy-induced hypertension
* more than 2 cesarean sections in patient's medical history
* significantly increased risk of obstetric hemorrhage (placenta previa)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Adequacy of spinal anesthesia | 60min
  Level of surgical anesthesia at least T5 and no need for additional intraoperative analgesia

SECONDARY OUTCOMES:
Number of complications | 60min
  Hypotension, bradycardia, nausea, vomiting,
Postoperative opioid consumption | 24hours
  Time to the first dose of morphine and total amount of morphine used postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Malec-Milewska, MD, Study Chair — Centre of Postgraduate Medical Education
Locations (1):
- Centre of Postgraduate Medical Education,Department of Anesthesia and Intensive Care, Warsaw, Poland